CLINICAL TRIAL: NCT04220086
Title: The Effectiveness and Brain-related Mechanism of Pediatric Massage for Children With Autism Spectrum Disorder (ASD): A Randomized, Waiting-list Controlled Trial
Brief Title: Pediatric Massage for Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Shenzhen Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNASD1
Record Dates: First submitted 2019-10-27; First posted 2020-01-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pediatric massage (Experimental): Children with ASD will receive pediatric massage for 12 weeks.
  Interventions: Procedure: Pediatric massage therapy; Procedure: Usual care
- Waitlist control (Sham Comparator): Waitlist control
  Interventions: Procedure: Usual care
- Healthy Control (Other): 15 healthy controls (age- and sex- matched with ASD patients) will be recruited. All of them will receive clinical evaluations, EEG and fNIRS detection.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Pediatric massage therapy — Children with ASD will receive pediatric massage therapy twice a week for 12 consecutive weeks by professional pediatric massage doctor. In addition, they will receive parent provided pediatric massage therapy at home after their parents received the professional pediatric massage therapy training. The frequency of pediatric massage will not be more than once every day and each session last about 30 minutes.
  Arms: Pediatric massage
Procedure: Usual care — Including Applied Behavior Analysis (ABA), Educational intervention, Interpersonal development intervention.
  Arms: Pediatric massage; Waitlist control
Other: No intervention — No intervention for healthy controls
  Other Names: No intervention for healthy controls
  Arms: Healthy Control

SUMMARY:
This study was designed as a randomized controlled clinical trial of pediatric massage for children with Autism Spectrum Disorder (ASD). 72 ASD children will be recruited and randomly divided into two groups: the treatment group (pediatric massage + usual care, n=36) and the control group (usual care/waitlist group, n=36).30 healty controls will be recruited. Children in the treatment group will received 12 weeks pediatric massage by doctors and their own parents.

The Autism Behavior Checklist (ABC), Childhood Autism Rating Scale (CARS), Autism Treatment Evaluation Checklist (ATEC), Social Responsiveness Scale-Second Edition (SRS-2), Children's Sleep Habits Questionnaire (CSHQ) and Eysenck Personality Questionnaire (EPQ) will be used to assess the clinical behavioral changes of all participants, and to analyze the clinical effectiveness and safety of pediatric massage for children with ASD.

Electroencephalography (EEG) and brain functional near-infrared spectroscopy (fNIRS) will be recorded before and after treatment, to observe the potential brain target of pediatric massage for children with ASD.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by deﬁcits in social interactions and communication skills, both verbal and non-verbal, restricted interests, and stereotypical behaviors. However, at present, there is no drug has proven effective in alleviating the core symptoms of social and communication difficulties in ASD.

ASD families are becoming turn to complementary and alternative medicine (CAM). They use CAM to treat symptoms of autism in general, comorbid symptoms (such as attention, hyperactivity, irritability, moodiness, gastrointestinal symptoms, seizures, sleep and tactile sensitivity). In addition, some families report that the use of CAM has less negative side effects compared with conventional treatments.

As a traditional TCM therapy, pediatric massage has been used in treating various pediatric diseases including ASD. A large number of clinical studies have shown that pediatric massage can improve ASD and its accompanied symptoms effectively. However, its exact effectiveness and mechanism need to be further explored.

In the proposed study, pediatric massage will be employed to treat children with ASD, to confirm the effectiveness and safety of pediatric massage therapy for children with ASD, and to explore the potential mechanism and target of pediatric massage for ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Autism Spectrum Disorder (ASD) has been diagnosed and a diagnosis certificate has been provided. The diagnostic criteria is based on the Diagnostic and Statistical Manual of Mental Disorders fifth version (DSM-V) criteria of Autism Spectrum Disorder. Score of CARS≥30;
2. Aged 3-10, right-handedness ；
3. The parents (or other legal guardians) of participants to give consent and to cooperate with the treatment and data collection.

Exclusion Criteria:

1. The conventional treatment accepted currently does not belong to the following three categories: Applied Behavior Analysis (ABA), Educational intervention or Interpersonal development intervention;
2. Patients with any major treatment changes within 4 weeks prior to joining the study;
3. Patients or their parents with other neurodevelopmental disorders, severe psychiatric diseases, genetic disease, or other severe systemic disease (such as history of severe head trauma, or stroke);
4. Seizure within the last year prior to enrolment, or the need for seizure medications either at present or in the past;
5. Being involved in other clinical trials;
6. Patients received pediatric massage therapy in the past two months, or are receiving pediatric massage;
7. During the study period, parents will be required not to initiate any new interventions or modify current interventions unless absolutely necessary. If a change must be made, the parent is required to inform investigator, who decides whether the subject should stop participating in the study based on situation.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Autism Behavior Checklist (ABC) | Baseline, 4 week, 8 week, 12 week, and follow-up assessment at the week of 4, 8, 12 after treatment
  ABC is a scale used for nonadaptive behaviors created to screen and indicate the probability of a diagnosis of autism. The questionnaire including 57 items related to five areas: sensorial, relational, use of body and objects, and social skills. Scale score> 67 strongly suggests the presence of autism. Changes in the ABC from baseline to endpoint will be observed. Assessments will be conducted at baseline and once every four weeks thereafter.

SECONDARY OUTCOMES:
Changes in the Childhood Autism Rating Scale (CARS) | Baseline, 4 week, 8 week, 12 week
  CARS assesses the child on a scale from 1 to 4 in each of 15 dimensions or symptoms (including the ability to relate to people, emotional response, imitation, body use, object use, listening response, fear or nervousness, verbal communication, nonverbal communication, activity level, level and reliability of intellectual response, adaptation to changes, visual response, taste, smell and touch responses and general impressions). A total score of at least 30 strongly suggests the presence of autism. Children with score between 30 and 36 have mild-to-moderate autism while those with score between 37 and 60 have severe autism. Change in CARS from Baseline to Endpoint will be observed. Assessments will be conducted at baseline and once every four weeks thereafter.
Changes in the Social Responsiveness Scale - Second Edition (SRS-2) | Baseline, 4 week, 8 week, 12 week
  The Social Responsiveness Scale is a parent- and/or teacher-reported 65 question scale designed to measure social competence. Each question on the scale inquires about an observed aspect of reciprocal social behavior that is rated from "0" to "3", where 0 is best possible behavior and 3 is the worst possible behavior. The total SRS score may range from 0 to 195 where higher values represent the worse outcome. Assessments will be conducted at baseline and once every four weeks thereafter.
Changes in the Children's Sleep Habits Questionnaire (CSHQ) | Baseline, 4 week, 8 week, 12 week
  The Children's Sleep Habits Questionnaire (CSHQ) is a parental report sleep screening instrument designed for preschool- and school-aged children. The scale yields both a total score and 8 subscales reflecting the following sleep domains:1) bedtime resistance, 2) sleep onset delay, 3) sleep duration, 4) sleep anxiety, 5) night wakings, 6) parasomnias, 7) sleep-disordered breathing, 8) daytime sleepiness. Each item is answered with 1 of 3 markers: "usually" for 5 or more times a week, "sometimes" for 2-4 times a week, and "rarely" for never or 1 time a week. Higher scores reflect more disturbed sleep behavior. Assessments will be conducted at baseline and once every four weeks thereafter.
Changes in the Eysenck Personality Questionnaire (EPQ) - adult version | Baseline
  The EPQ is a three dimensional personality assessment tool to assess the personality traits of a person, including the Psychoticism (P), Extraversion (E), Neuroticism (N), and Lie (L) scales. Assessments will be conducted at baseline for parents to access parents' personality.
Changes in electroencephalography (EEG) | Baseline, 12 week
  EEG is a useful indicator of cortical connectivity between functional areas in the brain. Continuous resting-state electroencephalography (EEG) was recorded before and after the 12-week treatment and the delta (δ), theta (θ), alpha (α), beta (β) and gamma (γ) bands frequency will be used for EEG analysis.
Changes in functional near-infrared spectroscopy (fNIRS) of the brain | Baseline, 12 week
  Functional near-infrared spectroscopy (fNIRS) is a non-invasive neuroimaging procedure used to measure hemodynamic changes (oxyhemoglobin, deoxyhemoglobin and total haemoglobin), it will be measured at baseline and after the12-week treatment.
Number of participants with non-serious and serious adverse events (AEs) | 1,2,3,4,5,6,7,8,9,10,11,12 weeks
  Safety assessment. Adverse events that are related to treatment will be recorded once AE happens throughout the whole study. Adverse events rate will be assessed in all patients.
Number of participants with abnormal laboratory values in blood routine examination. | Baseline, 12 week
  Safety assessment. Blood routine examination (including RBC, WBC, Hb, HCT, PLT, MCV, MCH, MCHC, W-SCR, W-LCR, W-SCC, W-LCC, RDW-CV, PDW, and MPV levels) will be conducted before and after treatment to evaluate if there is infection or anemia. Number of participants with abnormal laboratory values will be recorded.
Changes in the Autism Treatment Evaluation Checklist (ATEC). | Baseline, 4 week, 8 week, 12 week
  The ATEC is designed to be completed by parents, teachers, or caretakers. It consists of 4 subtests: I. Speech/Language Communication (14 items); II. Sociability (20 items); III. Sensory/ Cognitive Awareness (18 items); and IV. Health/Physical/Behavior (25 items). It basically provides several subscale scores as well as a total score to be used for comparison before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, Principal Investigator — The University of Hong Kong-Shenzhen Hospital
Locations (2):
- China (2):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Department of Chinese Medicine, The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided